CLINICAL TRIAL: NCT05773170
Title: Retrospective Registry for the Efficacy and Safety Evaluation of Refralon®, Concentrate for Solution for Intravenous Injection in Patients With Paroxysmal and Persistent Atrial Fibrillation and Flutter
Brief Title: Efficacy and Safety Evaluation of Refralon®, Concentrate for Solution for Intravenous Injection in Patients With Paroxysmal and Persistent Atrial Fibrillation and Flutter
Status: Completed | Type: Observational
Sponsor: R-Pharm (Industry)
Collaborators: FSBI "National Medical Research Center of Cardiology named after academician E.I.Chazov" of the Ministry of Health of the Russian Federation (Unknown)
Responsible Party: Sponsor
Other Study IDs: CC01897112
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation; Atrial Flutter
Keywords: pharmacological cardioversion; antiarrhythmic; intravenous administration; paroxysmal and persistent atrial fibrillation and flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pharmacological cardioversion with Refralon: 1. Refralon® 0.1% solution administration at a dose of 10 μg/kg of body weight intravenously (IV) for 2-3 minutes; It is allowed to divide the first Refralon® bolus into two consecutive injections: the first dose administration - 5 μg/kg of body weight, if the AF/AFL persists, administer the second dose - 5 μg/kg of body weight (total dose 10 μg/kg) in 15 minutes.
  2. If no effect is registered (no sinus rhythm restoration), repeat IV administration of Refralon® 0.1% solution at a dose of 10 μg/kg of body weight (total dose: 20 μg/kg of body weight) in 15 minutes;
  3. If no effect is registered, repeat IV administration of Refralon® 0.1% solution at a dose of 10 μg/kg of body weight (total dose: 30 μg/kg of body weight) in 15 minutes.
  In case of AF/AFL recurrence after the sinus rhythm restoration (with no contraindications), it is possible to re-administer Refralon®, while the maximum total drug daily dose (from the first administration) should not exceed 30 μg/kg of body weight.
  Interventions: Drug: Refralon

INTERVENTIONS:
Drug: Refralon — 1 mg/ml concentrate for solution for intravenous injection. (Prior to the administration, 2 mL of Refralon® must be diluted to 20 mL in 0.9 % sodium chloride).
  Other Names: 4-nitro-N-[(1RS)-1-(4-fluorophenyl)-2-(1-ethylpiperidin-4-yl)ethyl]benzamide hydrochloride; Niferidyl

SUMMARY:
The goal of this retrospective registry is to evaluate the efficacy and safety of Refralon®, concentrate for solution for intravenous injection, as chemical cardioversion in patients with paroxysmal and persistent atrial fibrillation and flutter in routine clinical practice. The main questions it aims to answer are:

* What is the incidence of sinus rhythm restoration within 6 hours in patients with paroxysmal atrial fibrillation (AF)/atrial flutter (AFL) after the first dose of Refralon®?
* What is the incidence of sinus rhythm restoration within 24 hours in patients with persistent AF/AFL after the first dose of Refralon®?

DETAILED DESCRIPTION:
The registry is a retrospective multicenter observational study in patients with paroxysmal and persistent forms of AF and AFL who underwent chemical cardioversion with Refralon® in a hospital setting.

After the compliance with the inclusion criteria and the absence of exclusion criteria based on medical documentation, the patient data will be collected from medical documentation available for the analysis into a unified electronic case report form (eCRF).

Alongside the study therapy, all the patients must receive an adequate anticoagulant therapy in accordance with the current clinical guidelines of the Ministry of Health of the Russian Federation. After chemical cardioversion, patients were followed up and examined as a part of routine clinical practice. The examination data will be used for this study analysis. No additional therapeutic or diagnostic procedures are provided by the analysis protocol.

Study patient follow-up period was 24 hours from the Refralon® first dose administration.

The patients' data collection is planned for 8 months. It is planned to enroll 1500 patients with persistent and paroxysmal AF and AFL, meeting the inclusion/exclusion criteria. If necessary, it is possible to extend the registry data collection period to include the planned number of patients.

Approximately in 3 and 6 months from the registry initiation (but not earlier than after the inclusion of 150 patients into the registry), an interim collected data analysis can be performed in order to preliminary assess the Refralon® efficacy and safety data in this study, as well as to identify the potential data entry errors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: paroxysmal or persistent atrial fibrillation or flutter;
* A chemical cardioversion procedure performed with Refralon® in a hospital setting.

Exclusion Criteria:

* Congenital or acquired QT interval prolongation in the electrocardiogram (ECG) in 12 standard leads for more than 440 ms at the time of cardioversion;
* Bradysystolic atrial fibrillation or flutter (mean heart rate < 50 bpm or pauses > 3 sec, registered on the ECG or identified by the results of 24-hour Holter ECG monitoring, except for the cases of its correction by a cardiac pacemaker at the time of cardioversion;
* Sick sinus syndrome (sinus bradycardia, sinoatrial blockade), previously registered as associated with sinus rhythm, except for the cases of its correction with a cardiac pacemaker at the time of cardioversion;
* Degree II - III atrioventricular blockade, two- and three-beam blockade with no cardiac pacemaker at the time of cardioversion;
* Acute myocardial infarction period at the time of cardioversion;
* Acute period after coronary artery bypass grafting (CABG) or other cardiac surgery (at least 7 days after CABG at the time of cardioversion);
* Decompensated or severe chronic heart failure (III-IV functional class according to New York Heart Association (NYHA) classification) at the time of cardioversion;
* Uncontrolled bronchial asthma, severe respiratory failure at the time of cardioversion;
* Pregnancy and breastfeeding at the time of cardioversion;
* Administration of Class IA antiarrhythmic drugs (quinidine, hydroquinidine, disopyramide, procainamide) at the time of cardioversion;
* Class III antiarrhythmic drugs administration at the time of cardioversion;
* Cardiac glycosides administration at the time of cardioversion;
* Administration of QT-prolonging drugs at the time of cardioversion;
* Heart rate < 50 bpm, pauses > 3 seconds on the ECG or Holter ECG monitoring (HM-ECG) during wakefulness at the time of cardioversion;
* Hyperthyroidism or decompensated hypothyroidism (thyroid stimulating hormone (TSH) < lower limit of normal or > 2 upper limits of normal) at the time of cardioversion;
* Uncorrectable electrolyte disorders (potassium level less than 3.5 mmol/L) at the time of cardioversion;
* Identified contraindications to the sinus rhythm restoration at the time of cardioversion;
* Blood clots in the heart cavities or spontaneous grade III-IV echo contrast at the time of cardioversion according to transesophageal echocardiography;
* The need for electrical cardioversion due to the patient's hemodynamic instability at the time of cardioversion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patient cohort with paroxysmal and persistent AF and AFL who underwent chemical cardioversion with Refralon®, concentrate for solution for intravenous injection, in accordance with the patient information leaflet, the current clinical guidelines of the Ministry of Health of the Russian Federation, and the approved treatment standards for AF and AFL patients in the clinical centers.
Sampling Method: Non-Probability Sample
Enrollment: 1147 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of sinus rhythm restoration | up to 6 hours
  Incidence of sinus rhythm restoration within 6 hours in patients with paroxysmal AF/AFL after the first dose of Refralon®
Incidence of sinus rhythm restoration | up to 24 hours
  Incidence of sinus rhythm restoration within 24 hours in patients with persistent AF/AFL after the first dose of Refralon®

SECONDARY OUTCOMES:
Time from the Refralon® administration start to the sinus rhythm restoration | from Refralon® administration to the sinus rhythm restoration, up to 24 hours
Incidence of sinus rhythm maintenance | up to 24 hours
  Incidence of sinus rhythm maintenance in patients 24 hours after the first Refralon® dose
Incidence of AF/AFL sustained recurrences | up to 24 hours
  Incidence of AF/AFL sustained (for more than 30 seconds) recurrences within 24 hours after the successful cardioversion with Refralon®

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — Chief Medical Officer, R-Pharm
Locations (33):
- Russia (33):
  - Federal State Budgetary Educational Institution of Higher Education "Bashkir State Medical University" of the Ministry for Healthcare of the Russian Federation, Ufa, Bashkortostan Republic
  - State Budgetary Healthcare Institution of Republic of Bashkortostan "City Hospital Clinical Hospital № 21", Ufa, Bashkortostan Republic
  - State Autonomous Healthcare Institution of the Kemerovo Region "Novokuznetsk City Clinical Hospital № 1", Novokuznetsk, Kemerovo Oblast
  - State Budgetary Healthcare Institution of Sverdlovsk Region "Scientific-practical center of specialized typed of medical care "URAL INSTITUTE OF CARDIOLOGY", Yekaterinburg, Sverdlovsk Oblast
  - "First Clinical Medical Center" LLC, Kovrov, Vladimirskaya Oblast’
  - The Regional State Budgetary Healthcare Institution "St. Joseph Belgorod Regional Clinical Hospital", Belgorod
  - State budgetary Healthcare Institution "Cardiological Dispensary", Ivanovo
  - Federal State Budgetary Institution "National Medical Research Center for Therapy and Preventive Medicine" of the Ministry of Healthсare of the Russian Federation, Moscow
  - State Budgetary Healthcare Institution "City Clinical Hospital named after I.V. Davydovsky of Moscow Healthcare Department", Moscow
  - Federal State Budgetary Institution "Clinical hospital № 1" administrative Department of the President of the Russian Federation, Moscow
  - Federal State Budget Institution "A.N. Bakulev National Medical Research Center of Cardiovascular Surgery" of the Ministry of Health of the Russian Federation, Moscow
  - State Budgetary Healthcare Institution of the Novosibirsk Region "Novosibirsk Regional Clinical Cardiology Dispensary", Novosibirsk
  - State Budgetary Healthcare Institution of the Novosibirsk region "City Clinical Hospital № 2", Novosibirsk
  - Clinical Health Unit No. 9, Omsk
  - State Budgetary Healthcare Institution of the Perm Region "Clinical Cardiological Dispensary, Perm
  - State Budgetary Institution of the Ryazan region "Regional Clinical Cardiology Dispensary", Ryazan
  - St. Petersburg State Budgetary Healthcare Institution "Hospital for War Veterans", Saint Petersburg
  - Federal State Budgetary Institution "National Medical Research Center (NMIC) named after V. A. Almazov" Ministry of Health Russia, Saint Petersburg
  - The Saint Petersburg State Health Care Establishment the City Hospital № 40 of the Resort District, Saint Petersburg
  - The State Budgetary Healthcare Institution of the Samara Region "Samara Regional Clinical Cardiology Dispensary named after V.P. Polyakov", Samara
  - Samara City Clinical Hospital № 1 named after N.I. Pirogov, Samara
  - State Health Care Institution "Regional Cardiology Clinic", Saratov
  - Tambov Regional State Budgetary Healthcare Institution "S.S. Bryukhonenko City Hospital of Michurinsk", Tambov
  - Cardiology Research Institute, Federal State Budgetary Scientific Institution "Tomsk National Research Medical Center of the Russian Academy of Sciences", Tomsk
  - State health institution City Hospital № 13 Tula (Tula regional cardiological dispensary), Tula
  - The State Budgetary Healthcare Institution of the Tver region "Regional Clinical Hospital", Tver'
  - The State Budgetary Healthcare Institution of the Vladimir Region "State Hospital № 4", Vladimir
  - The State Budgetary Healthcare Institution "Volgograd Regional Clinical Cardiology Center", Volgograd
  - Budget Healthcare Institution of the Vologda Region "Vologda Regional Clinical Hospital", Vologda
  - The State Healthcare Institution "Voronezh Regional Hospital № 1", Voronezh
  - The State Budgetary Health Care Institution of the Yaroslavl Region "Regional Clinical Hospital", Yaroslavl
  - State Budgetary Healthcare Institution "Sakhalin Regional Clinical Hospital", Yuzhno-Sakhalinsk
  - State Budgetary Healthcare Institution of the Sakhalin region "Yuzhno-Sakhalinsk City Hospital named after F.S. Ankudinov", Yuzhno-Sakhalinsk